CLINICAL TRIAL: NCT03502824
Title: A Prospective, Multicenter, Randomized, Controlled Clinical Study Of PuraPly® AM and Standard of Care (SOC) Compared to SOC Alone For The Management Of Stage II-IV Pressure Ulcers
Brief Title: PuraPly® AM Plus the Standard of Care to Standard of Care Alone for the Management of Stage II-IV Pressure Ulcers.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow enrollment
Sponsor: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-PRU-004-PPAM
Record Dates: First submitted 2018-04-09; First posted 2018-04-19 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Chronic Pressure Ulcers
Keywords: Chronic wounds; PHMB; Pressure Ulcer; Wound Management; Collagen; Stage II; Stage III; Stage IV; Pressure Injury
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PuraPly® AM plus Standard of Care (Active Comparator)
  Interventions: Device: PuraPly® Antimicrobial Wound Matrix
- Standard of Care (SOC) for Pressure Ulcers (Active Comparator)
  Interventions: Other: SOC for Pressure Ulcers

INTERVENTIONS:
Device: PuraPly® Antimicrobial Wound Matrix — PuraPly® AM is a class II medical device, that has been 510(k) cleared by US Food and Drug Administration (FDA) (K051647) and is intended for the management of acute and chronic wound management across a variety of wound types, including partial- and full-thickness wounds, pressure ulcers, surgical wounds, trauma wounds, venous and diabetic ulcers.
  Other Names: PuraPly® AM
  Arms: PuraPly® AM plus Standard of Care
Other: SOC for Pressure Ulcers — SOC group will receive institutional standard of care which includes, but is not limited to, debridement, negative pressure wound therapy (i.e. VAC), ensuring perfusion and oxygenation, evaluating nutritional status and addressing deficits, offloading, keeping the ulcer bed moist with appropriate cleansing at the time of each dressing change. Standard dressings may include hydrocolloids, alginates, transparent film, foam, moist gauze dressings. In addition, a non-toxic topical antiseptic, may be used per NPUAP Clinical Practice Guidelines (2014) for SOC group only, if colonization is suspected.
  Arms: Standard of Care (SOC) for Pressure Ulcers

SUMMARY:
This is a prospective, multi-center, randomized, controlled clinical study Of PuraPly® AM and standard of care (SOC) compared to SOC alone for the management of Stage II-IV pressure ulcers located in the gluteal, ischial, hip, sacral, coccygeal, and trochanteric, malleolus, or heel area.

DETAILED DESCRIPTION:
This study seeks to demonstrate how PuraPly® AM performs against standard of care in Stage II-IV Pressure Ulcers through a prospective randomized controlled study design.

Subjects may be enrolled for up to 24 weeks; if healing occurs prior to week 24, a follow up healing confirmation visit shall occur two weeks later to confirm maintenance of complete wound closure and participation may continue up to 24 weeks. Subjects that are randomized to the SOC group have the opportunity to cross over and receive PuraPly AM at week 12 if their index ulcer has not healed; they will then be followed for an additional 12 weeks for up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. Subject has a Stage II-IV pressure ulcer located in the gluteal, ischial, hip, sacral, coccygeal, and trochanteric, malleolus, or heel area.
3. Pressure ulcer should be present for 4 weeks duration and have a ulcer surface area > 2cm2
4. If multiple ulcers are present, one ulcer must be identified as the index ulcer.
5. The index ulcer is free from active infection at the time of randomization.
6. Willingness to off-load or pressure redistribute ulcer for duration of enrollment
7. The index ulcer has been offloaded for at least 7 days prior to randomization.
8. The index ulcer must have been present for at least 30 days at time of study enrollment.
9. The index ulcer is separated at least 4 cm from all other ulcers at Study Day -7 and Study Day 0 (post-debridement) and has a margin of intact skin sufficient for anchoring of the required study dressing.
10. Subject has read and signed the IRB/IEC approved Informed Consent Form (ICF) before screening procedures are undertaken.

Exclusion Criteria:

1. Presence of signs and symptoms of infection at the index ulcer site, including but not limited to cellulitis, acute osteomyelitis, excessive exudate, gangrene or deep tissue infection
2. The index ulcer is not free of necrotic tissue and is unable to tolerate debridement
3. Non-enteric or unexplored sinus tract
4. Concomitant conditions that in the judgment of the investigator would make the subject inappropriate for entry to the study
5. Subject has a known sensitivity to porcine materials
6. Subject has a known sensitivity to polyhexamethylenebiguanide (PHMB)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Reduction in size of ulcer area between groups | Up to 24 weeks
  As measured from change in size from baseline
Improvement in wound bed condition between groups | Up to 24 weeks
  As measured from change in status from baseline

SECONDARY OUTCOMES:
Time to complete wound closure between both groups | Up to 24 weeks
  As measured by time to complete wound closure from baseline
Improvement in patient reported pain | Up to 24 weeks
  As measured change in status from baseline as assessed by the PAIN visual analogue scale (PAIN-VAS)
Improvement in patient reported quality of life | Up to 24 weeks
  As measured by change in status from baseline as assessed by the Wound QoL (W-QoL), questionnaire on quality of life with chronic wounds

CONTACTS AND LOCATIONS:
Overall Officials: Scott Gorenstein, MD FACEP, Principal Investigator — NYU Winthrop Hospital; Alisha Oropallo, MD, FACS, APWCA, Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Northwell Health, Lake Success, New York
  - NYU Winthrop Hospital, Mineola, New York

IPD SHARING:
Plan to Share IPD: Undecided